CLINICAL TRIAL: NCT00731302
Title: Vascular Damage in Systemic Lupus Erythematosus (SLE)
Brief Title: Aspirin Resistance in Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine, Professor of Pharmacology, Associate Director of the Division of Clinical Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HL65082; R01HL065082 (NIH)
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Aspirin; Meloxicam; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aspirin and Meloxicam (Experimental): Arm: Aspirin and Meloxicam Each participant will receive 81 mg aspirin per day for 7 days, followed by meloxicam 7.5 mg daily plus aspirin 81 mg daily for 5 days
  Interventions: Drug: aspirin and meloxicam

INTERVENTIONS:
Drug: aspirin and meloxicam — aspirin 81 mg daily then aspirin 81 mg plus meloxicam 7.5 mg daily
  Other Names: generic, not applicable

SUMMARY:
This study examine whether patients with lupus respond to aspirin , and if not, if that is related to inflammation. We examine the ability of aspirin to inhibit the production of thromboxane in patients with lupus and controls and see if aspirin insensitive thromboxane production is inhibited by meloxicam.

DETAILED DESCRIPTION:
Premature cardiovascular disease is a major cause of mortality in patients with systemic lupus erythematosus (SLE) with the risk of myocardial infarction increased up to 50-fold. In addition to defining the mechanisms for accelerated atherosclerosis it is important to define the effects of drugs used to reduce cardiovascular risk in high-risk patients. Low dose aspirin, by inhibiting thromboxane A2 biosynthesis, has profound antiplatelet effects, but some patients have impaired thromboxane suppression - a phenomenon termed aspirin resistance. An explanation is that aspirin-independent thromboxane synthesis may occur through enhanced COX-2 activity, as would occur in an inflammatory condition such as lupus. However, little is known about the effects of low-dose aspirin in SLE. Thus, we propose to test the following hypothesis: 1) that aspirin insensitive thromboxane biosynthesis is increased in patients with lupus and is mediated by increased COX-2 activity.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent.
* Age >18 yrs.
* SLE meeting ACR criteria {Tan, Cohen, et al. 1982 1482 /id} for at least 6 months.(SLE group)
* Stable disease activity as evidenced by no change in immunosuppressive therapy in the past 1 month.
* If female of childbearing potential must use an effective method of birth control

Exclusion criteria.

* Renal disease (creatinine >1.5 mg/dL, dialysis, 2+ or more proteinuria)
* Previous or current history of peptic ulcer disease or gastrointestinal bleed.
* Previous or current thromboembolic or ischemic cardiovascular event (stroke, myocardial infarction, angina) - can do aspirin part of study.
* Currently taking an anticoagulant or antiplatelet agent (besides aspirin).
* Thrombocytopenia (platelet count <135,000)
* Pregnancy
* Allergy to aspirin, NSAIDs
* NSAIDs in the previous week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
thromboxane | after aspirin and after aspirin plus meloxicam
  a hormone of the prostacyclin type released from blood platelets. It induces platelet aggregation and arterial constriction.

CONTACTS AND LOCATIONS:
Overall Officials: C M Stein, M.D., Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Vanderbilt University Medical School, Nashville, Tennessee

REFERENCES:
- [Result] Kawai VK, Avalos I, Oeser A, Oates JA, Milne GL, Solus JF, Chung CP, Stein CM. Suboptimal inhibition of platelet cyclooxygenase 1 by aspirin in systemic lupus erythematosus: association with metabolic syndrome. Arthritis Care Res (Hoboken). 2014 Feb;66(2):285-92. doi: 10.1002/acr.22169. PMID 24022862